CLINICAL TRIAL: NCT06309771
Title: Influence of a Complex Behavioural Intervention on the Quality of Life of Medical Students: A Randomized, Controlled, Single-Center Study.
Brief Title: Preventive Remediation for Optimal MEdical StudentS (PROMESS)
Acronym: PROMESS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Research on Healthcare Performance Lab U1290 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PROMESS - QOL
Record Dates: First submitted 2023-11-08; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Health Behavior; Health-Related Behavior
Keywords: Health; Student; Curriculum; Behavior; Quality of life; Medical; Performance; Stress; Sleep; Fatigue; Sedentary behaviors; Physical Activity; Medical pedagogy
MeSH Terms: conditions — Health Behavior; Behavior; Fatigue; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial. Randomization into two groups: INTERVENTION group and CONTROL group. The INTERVENTION group will have the opportunity to follow a preventive remediation program based on 3 modules: stress management, sleep improvement and fatigue reduction, and sedentary behaviors reduction and physical activity promotion. The order of following the 3 modules will be randomized. The CONTROL group will not receive any intervention.
Who Masked: Outcomes Assessor
Masking Description: Assessors of pre and posttest measures will be blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Complex behavioral intervention based on health-related modules.
  Interventions: Behavioral: Stress management, sleep improvement and fatigue reduction, sedentary behaviors reduction and physical activity promotion.
- Control (No Intervention): Students from the control group will follow no modules.

INTERVENTIONS:
Behavioral: Stress management, sleep improvement and fatigue reduction, sedentary behaviors reduction and physical activity promotion. — The study seeks to quantify the impact of a complex intervention based on 3 modules :
  1. Stress management
  2. Sleep improvement and fatigue reduction,
  3. Sedentary behaviors reduction and physical activity promotion.
  Students from the interventional group will follow these 3 different health-related modules in a random order (6 predetermined order). Each module will be composed on 3 sessions. Each session includes individual interviews covering initial assessment and personalized goal setting.
  Arms: Intervention

SUMMARY:
Medical students are under a great deal of competitive pressure throughout their training. During their studies, medical students experience high levels of stress, sleep disorders and excessive physical inactivity. These feelings and behaviours are expected to significantly degrade their quality of life, health and performance.

The PROMESS project aims to increase students' quality of life and ultimately improve their medical performance. The project aims to improve students' ability to take care of themselves from a short and long term perspective.

Encouraging physical activity, reducing sedentary behaviors, reducing stress, fatigue and sleep troubles during their curriculum can promote a healthier lifestyle and reduce the risk of chronic health conditions in the future.

The study seeks to quantify the impact of a complex intervention based on 3 modules (stress, sleep, physical activity) on the quality of life and academic performance of 2nd cycle medical students. This study will also have a clear insight on the influence of the complex intervention on changes in stress, sleep, physical activity and sedentary behavior markers.

DETAILED DESCRIPTION:
Our project aims to help future healthcare professionals to adopt health-promoting behaviors during their studies in a preventive approach. This support will be provided through a multimodal intervention during their curriculum. Specifically, 4th and 5th-year students at the Faculty of Medicine of Lyon Est will have the opportunity to participate in the PROMESS project. Voluntary will be randomized into 2 arms (intervention and control). The control group will not receive any intervention. The intervention group will follow a preventive program based on three modules: sedentary behaviors reduction and physical activity promotion, stress management, and sleep improvement and fatigue reduction. This program will span 30 weeks. Both groups will be characterized through a pre- post paradigm multimodal measurement. At the end of this period, we expect improvements in terms of quality of life, physical and mental health, and performance in the interventional arm.

METHODS.

POPULATION. The population consists of 70 medical students, with 2/3 (n=45 students) assigned to the intervention group and 1/3 (n=25 students) to the control group.

PRE-INTERVENTION. From week 1 to 3. All students will undergo a two-hour session, during which, they will complete questionnaires on sedentary behavior and physical activity, stress, sleep and fatigue levels. Bioimpedance and Heart Rate Variability will be measure. Students will perform three physical fitness tests (vertical jump, maximal isometric strength, and endurance). Then, they will wear actimeters to record sleep, sedentary behaviors and physical activity levels during three weeks.

INTERVENTION. From week 5 to week 25. The intervention program aims to address three key aspects of well-being. The students in the intervention group will take part in three modules, one on stress, one on sleep and fatigue, and the other on sedentary behaviors and physical activity.

The order of the 3 modules will be randomized so that each student will perform a specific module during one phase (e.g., a student will undergo the sleep module during the first phase, the stress module during the second phase, and the physical activity module during the third phase). Each module will consist of three individual sessions, each lasting one hour, with approximately 15 days between each session. Each session includes individual interview between an expert and the participant (i.e.student). The sessions will be scheduled as follow:

* First phase: week 5 and 6 (session 1), week 7 and 8 (session 2), week 9, 10, and 11 (session 3).
* Second phase: week 12 and 13 (session 1), week 14 and 15 (session 2), week 16, 17, and 18 (session 3).
* Third phase: week 19 and 20 (session 1), week 21 and 22 (session 2), week 23, 24, and 25 (session 3).

During the interview, the expert will realize an initial assessment of student health behaviors and will give personalized goals to student. Subsequent sessions follow the same structure. Subjective and objective indicators related to each intervention domain will be recorded to assess the progress of student.

DURING THE INTERVENTION. Week 1,4,7,10,13,16,19,22,25,28,30. Evolutionary monitoring with multi-dimensional Visual Analogues Scales (quality of life, stress, fatigue, sleep, sedentary behaviors, physical activity) for intervention and control groups.

POST-INTERVENTION. From week 27 to 29. All students will undergo the exact same set of measurements as described in pre-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Being a 4th-year or a 5th-year medical student at the Faculty of Medicine Lyon East during the academic year 2023-2024.
* Having read the information note.
* Having signed the written consent.

Exclusion Criteria:

* No exclusion criteria will be applied.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life. Change from pre-intervention in a composite score obtained at the Brief Quality Of Life questionnaire at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The students level of the quality of life is assessed four sub-scores of quality of life (i.e. physical health, psychic well-being, social relationship, environnement). The composite score is the mean of the 2 dimensions: physical health and psychological well-being.
  The measure will be done at different time frame:
  * Pre-intervention measure at week 1: before any involvement in the intervention (for the control and interventional groups).
  * Post-intervention measure at week 27 : after the intervention (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)

SECONDARY OUTCOMES:
Academic self-efficacy. Change from the pre-intervention in score obtained at the Academic self-efficacy questionnaire at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The students level of academic self-efficacy will be assessed through the Academic self-efficacy questionnaire ranging from 5 to 20. The measures will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the intervention (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the intervention (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Wu self efficacy questionnaire. Change from pre-intervention in score obtained at the adapted Wu self efficacy questionnaire at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The students level of self-efficacy will be assessed through the adapted Wu questionnaire ranging from 4 to 40. It can be divided into three sub-scores (i.e enrollment motivation, self-efficacy, learning engagement). The measures will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the intervention (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the intervention (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Academic performances. Scores and ranks obtained at all the official exams during the 2023-2024 academic year. | All along the project, in average 30 weeks.
  All the scores and ranks obtained at all the official exams during the 2023-2024 academic year will be recorded.
VAS - quality of life. Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) assessing the perceived level of Quality Of Life | Week 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 30
  The students level of the quality of life will be assessed on a 100-mm Visual Analogue Scale (VAS: "How would you describe your quality of life?") ranging from 0 (quality of life as bad as possible) to 100 (quality of life as good as possible).The measure will be done every 3 weeks from November to June in both groups, i.e. at week 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 30.
VAS - self-confidence. Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) assessing the perceived level of self-confidence. | Week 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 30
  The students level of self-confidence will be assessed on a 100-mm Visual Analogue Scale (VAS: "What is your self-confidence level?") ranging from 0 (No confidence at all) to 100 (Maximum confidence). The measure will be done every 3 weeks from November to June in both groups, i.e. at week 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 30
VAS - self-efficacy. Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) assessing the perceived level of self-efficacy. | Week 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 30
  The students level of the self-efficacy will be assessed on a 100-mm Visual Analogue Scale (VAS: "To what extent do you feel capable of succeeding in your student project?") ranging from 0 (Completely incapable) to 100 (Maximum capability). The measure will be done every 3 weeks from November to June in both groups, i.e. at week 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 30.
VAS - resources. Evolution of the score obtained at the 100-mm Visual Analogue Scale assessing the perceived level of resources. | Week 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 30
  The students level of resources will be assessed on a 100-mm Visual Analogue Scale (VAS: "Do you believe you have enough resources/tools at your disposal to succeed in your student project?") ranging from 0 (No, absolutely not) to 100 (Yes, completely). The measure will be done every 3 weeks from November to June in both groups, i.e. at week 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 30.
VAS - work-life balances. Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) assessing the work-life balances. | Week 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 30
  The work-life balances will be assessed on a 100-mm Visual Analogue Scale (VAS: "How would you rate your current work-life balance?") ranging from 0 (Completely unbalanced Work > Life) to 100 (Completely unbalanced Life > Work). The measure will be done every 3 weeks from November to June in both groups, i.e. at week 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 30.
VAS - stressors quantity. Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) assessing the perceived quantity of stressors. | Week 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 30
  The students quantity of stressors will be assessed on a 100-mm Visual Analogue Scale ((VAS: "In the past two weeks, how many stressful situations have you encountered?") ranging from 0 (maximum/extreme) to 100 (zero). The measure will be done every 3 weeks from November to June in both groups, i.e. at week 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 30.
VAS - stress quality: Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) assessing the emotional valence associated with the stress level. | Week 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 30
  The emotional valence associated of the students stress level will be assessed on a 100-mm Visual Analogue Scale (VAS: "Over the past two weeks, how would you characterize your stress?") ranging from 0 (very negative feelings) to 100 (very positive feelings). The measure will be done every 3 weeks from November to June in both groups, i.e. at week 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 30.
VAS - stress coping. Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) assessing the management of stressful situations. | Week 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 30
  The students management of stressful situations will be assessed on a 100-mm Visual Analogue Scale (VAS: "Over the past two weeks, how did you manage your stressful situations?") ranging from 0 (very bad stress coping) to 100 (excellent stress coping). The measure will be done every 3 weeks from November to June in both groups, i.e. at week 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 30.
VAS - stress quantity. Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) assessing the perceived level of stress. | Week 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 30
  The students level of stress will be assessed on a 100-mm Visual Analogue Scale (VAS: "Over the past two weeks, how would you characterize your stress level?") ranging from 0 (total absence of stress) to 100 (stress maximal). The measure will be done every 3 weeks from November to June in both groups, i.e. at week 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 30.
VAS - sleep quality. Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) characterizing the sleep quality. | Week 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 30
  The students level of sleep quality will be assessed on a 100-mm Visual Analogue Scale (VAS: "Over the past two weeks, how would you characterize your sleep?") ranging from 0 (the worst quality of sleep possible) to 100 (the best quality of sleep possible). The measure will be done every 3 weeks from November to June in both groups, i.e. at week 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 30.
VAS - sleep quantity. Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) assessing the quantity of sleep. | Week 1, 4, 7, 10, 13, 16, 19, 22, 25, 28
  The student level of sleep quantity will be assessed on a 100-mm Visual Analogue Scale (VAS: "Over the past two weeks, how would you characterize your sleep?") ranging from 0 (quantity of sleep largely insufficient) to 100 (quantity of sleep largely sufficient). The measure will be done every 3 weeks from November to June in both groups, i.e. at week 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 30.
VAS - sleep fatigue. Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) assessing the perceived level of fatigue. | Week 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 30
  The students level of fatigue will be assessed on a 100-mm Visual Analogue Scale (VAS: "Over the past two weeks, how would you characterize your physical and mental fatigue levels ?") ranging from 0 (extreme fatigue) to 100 (absence total of fatigue). The measure will be done every 3 weeks from November to June in both groups, i.e. at week 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 30.
VAS - physical fitness. Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) assessing the perceived level of physical fitness. | Week 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 30.
  The students level of physical fitness will be assessed on a 100-mm Visual Analogue Scale (VAS: "Over the past two weeks, how would you characterize your level of physical fitness?") ranging from 0 (bad shape) to 100 (best shape ever). The measure will be done every 3 weeks from November to June in both groups, i.e. at week 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 30.
VAS - physical activity. Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) assessing the level of physical activity. | Week 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 30.
  The students level of physical activity will be assessed on a 100-mm Visual Analogue Scale (VAS: "Over the past two weeks, how would you characterize your level of physical activity?") ranging from 0 (completely inactive) to 100 (extremely active). The measure will be done every 3 weeks from November to June in both groups, i.e. at week 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 30.
VAS - sedentary behaviors. Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) assessing the perceived level of sedentary behaviors. | Week 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 30.
  The students level of sedentary behaviors will be assessed on a 100-mm Visual Analogue Scale (VAS: "Over the past two weeks, how would you characterize your level of sedentary behaviors?") ranging from 0 (extremely sedentary) to 100 (absolutely not sedentary). The measure will be done every 3 weeks from November to June in both groups, i.e. at week 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 30.
Perceived level of stress. Change from pre-intervention in score obtained at the Perceived Stress Scale (PSS) at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The students level of stress will be assessed through the PSS questionnaire ranging from 0 (none) to 40 (extreme). One score is assessed and can be classified as low, moderate and elevated stress. The measures will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the intervention (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the intervention (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Coping strategies.Change from pre-intervention in scores obtained at the Brief Cope Inventory (BCI) at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The students coping strategies (social support, active resolution, positive thinking, and avoidance) will be assessed through the BCI questionnaire, each score ranging from 1 to 4; a high score indicating the behaviour was highly engaged. The measures will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Quantity of stressors. Score obtained at the Holmes and Rahe Questionnaire Inventory during the pre-intervention. | Week 1 (Pre-intervention).
  The quantity of stressors met by students during the last years will be assessed with the Holmes and Rahe Questionnaire inventory. One score is assessed and can be classified as low, medium and high risk of health degradation. This measure will be done during the pre-interventional period at week 1 (for the control and interventional groups).
Big-5. Scores obtained at the Big-5 questionnaire. | Week 1 (Pre-intervention).
  The students personality traits (i.e. agreeableness, openness, consciousness, extraversion, neuroticism) will be assessed through the Big-5 questionnaire. Each score ranges from one to five. This measure will be done during the pre-interventional period at week 1 (for the control and interventional groups).
Perceived level of sleep troubles. Change from pre-intervention in score obtained at the Pittsburgh Sleep Questionnaire Inventory (PSQI) at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The students level of sleep troubles will be assessed through the PSQI score ranging from 0 (none) to 21 (extreme). This score classified the presence or absence of sleep troubles. It can be divided into eight sub-scores (i.e., sleep quality, sleep latency, time spent in bed, sleep time, habitual sleep efficiency, sleep disturbance, use of sleeping medication and daytime dysfunction).
  The measure will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Epworth Sleepiness scale. Change from the pre-intervention in score obtained at the Epworth Sleepiness scale at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The students level of diurnal sleepiness will be assessed through the Epworth Sleepiness scale ranging from 0 (none) to 24 (extreme). The measures will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Multidimensional Fatigue. Change from the pre-intervention in score obtained at the Multidimensional Fatigue Inventory (MFI) at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The students level of fatigue will be assessed through the MFI questionnaire that covers various dimensions of fatigue, including general fatigue, physical fatigue, mental fatigue, reduced motivation, and reduced activity; ranging from 4 to 20. A total score can also be assessed (from 20 to 100). The measures will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Reduced composite scale of morningness. Score obtained at the reduced composite scale of morningness (RCSMS). | Week 1 (Pre-intervention)
  The students chronotype are assessed through the RCSMS. A total score can also be assessed (from 7 to 30). This measure will be done during the pre-interventional period at week 1 (for the control and interventional groups).
Perceived level of physical activity. Change from the pre-intervention in score obtained at the Global Physical Activity Questionnaire (GPAQ) at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The student level of physical activity will be assessed through the GPAQ questionnaire. Scores are expressed in MET.min week. It can be divided into six sub-scores (i.e. level of moderate and intense physical activity, physical activity during leisure activity, physical activity for locomotion, physical activity at work locomotion and sedentarity levels). The measures will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Perceived level of sedentary. Change from the pre-intervention in score obtained at the Rapid Physical Activity Questionnaire (RPAQ) at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The students level of sedentary will be assessed through the RPAQ questionnaire. This questionnaire includes questions about sedentary behaviors, such as time spent sitting down. Scores are expressed in hours per day for week and weekend days. The measures will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Heart rate variability (HRV) marker. Change from pre-intervention in cardiac coherence at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The students level of physiological stress will be assessed through the cardiac coherence, an HRV marker. The measures will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Heart rate variability (HRV) marker. Change from pre-intervention in the SDNN score in at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The students level of physiological stress will be assessed through the SDNN score, an HRV marker. SDNN is the standard deviation of the inter-beat-intervals (IBI) measured in ms, NN means "normal" beats, i.e, removing abnormal or false beats.The measures will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Heart rate variability (HRV) marker. Change from pre-intervention in the RMSSD score in at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The students level of physiological stress will be assessed through the RMSSD, an HRV marker. RMSSD is the most commonly measured form of HRV, it calculates the difference between successive inter-beat-intervals (IBI) in ms, squares these values and takes the root of the mean. The measures will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Heart rate variability (HRV) marker. Change from pre-intervention in the pnn50% score in at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The students level of physiological stress will be assessed through the pnn50%, an HRV marker. NN50 is the Number of pairs of successive intervals that differ by greater than 50ms. And pNN50 which is more typically used is the proportion of NN50 over all N-N intervals in a sample, expressed as a percentage.The measures will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Heart rate variability (HRV) markers.Change from pre-intervention in the Low frequency / High frequency ratio (LF/HF) ratio in at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The students level of physiological stress will be assessed through the LF/HF ratio, an HRV marker. The HF band is typically correlated with RMSSD and NN50, lower HF power is associated with stress and anxiety. It is primarily associated with activity in the parasympathetic nervous system. The LF band is typically associated with the sympathetic nervous system and the HF/LF ratio is often used as a measure of sympathetic-parasympathetic balance in the nervous system. The measures will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Actimetry records. Change from pre-intervention in Time in Bed at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The objective students level of sleep will be accessed through the actimetry recordings.The time in bed (in hours/day) refers to the total duration between the time an individual gets into bed with the intention of sleeping and the time he/she get out of bed. It includes both the time spent asleep (total sleep time) and any periods of wakefulness while in bed. Essentially, it represents the total time allocated for sleep, regardless of whether the individual is actually sleeping during that time. The measure will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Actimetry records. Change from pre-intervention in Total Sleep duration at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The objective students level of sleep will be accessed through the actimetry recordings. The total duration of sleep is obtained during a specified period, measured in hours/day. It represents the overall quantity of sleep obtained by an individual.The measure will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 sco
Actimetry records. Change from pre-intervention in Sleep efficiency at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The objective students level of sleep will be accessed through the actimetry recordings.The sleep efficiency is the ratio of total sleep time to the total time spent in bed, expressed as a percentage. It reflects how effectively one is sleeping during the time allotted for sleep. The measure will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Actimetry records. Change from pre-intervention in Sleep Onset Latency at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The objective students level of sleep will be accessed through the actimetry recordings. The sleep onset latency is the amount of time it takes for an individual to fall asleep after getting into bed, measured from the time the lights are turned off until sleep onset, reported in minutes.The measure will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Actimetry records. Change from pre-intervention in Wake after Sleep Onset at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The objective students level of sleep will be accessed through the actimetry recordings.The wake after sleep onset measures the total amount of time spent awake after initially falling asleep, reported in minutes. It reflects the disruptions in sleep continuity. The measure will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Actimetry records. Change from pre-intervention in Number of Awakenings at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The objective students level of sleep will be accessed through the actimetry recordings.The number of awakenings represents the frequency of brief awakenings during the sleep period. Each awakening may disrupt the continuity of sleep and impact sleep quality. The measure will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Actimetry records. Change from pre-intervention in Mid-sleep point at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The objective students level of sleep will be accessed through the actimetry recordings.The mid-sleep point refers to the midpoint of an individual's sleep period. It is calculated by finding the halfway point between the time of sleep onset (when the individual falls asleep) and the time of sleep offset (when the individual wakes up). The measure will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Actimetry records. Change from pre-intervention in Bedtime at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The objective students basal level of sleep will be accessed through the actimetry recordings. The bedtime is the time at which an individual goes to bed with the intention of sleeping.The measure will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Actimetry records. Change from pre-intervention in Sleep Onset time at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The objective students basal level of sleep will be accessed through the actimetry recordings.The sleep onset time refers to the time at which an individual falls asleep after initially getting into bed with the intention of sleeping, measured in minutes. The measure will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Actimetry records. Change from pre-intervention in Sleep Inertia at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The objective students basal level of sleep will be accessed through the actimetry recordings. The sleep inertia refers to the periods between wake-up time and get-up time, measured in minutes. The measure will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Actimetry records. Change from pre-intervention in Wake-up time at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The objective students basal level of sleep will be accessed through the actimetry recordings. The wake-up time refers to the time at which an individual awakens from sleep in the morning. The measure will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Actimetry records. Change from pre-intervention in Sleep regularity index at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The objective students basal level of sleep will be accessed through the actimetry recordings.The sleep regularity index is a measure that evaluates the consistency of an individual's sleep habits over a given period. It takes into account the regularity of bedtime and wake-up times on a daily basis. The higher the sleep regularity index, the more consistent and regular the individual's sleep habits are considered to be. The measure will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Actimetry records. Change from pre-intervention in Total activity at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The objective students levels of physical activity and sedentary behavior will be accessed through the actimetre recordings.The total activity time represents the total duration of physical activity within the monitoring period, measured in hours.The measure will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Actimetry records. Change from pre-intervention in Moderate-to-vigorous Physical Activity (MVPA) at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The objective students levels of physical activity and sedentary behavior will be accessed through the actimetry recordings. MVPA refers to physical activities that require moderate to high levels of effort and significantly increase heart rate and breathing. These activities contribute to improved cardiovascular health, fitness, and overall well-being. MVPA encompasses a range of activities that are more intense than sedentary behaviors but less intense than vigorous activities. MVPA is measured in minutes/day. The measure will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Actimetry records. Change from pre-intervention in light physical activity at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The objective students levels of physical activity and sedentary behavior will be accessed through the actimetry recordings. Light physical activity refers to any activity that requires minimal effort and only slightly elevated heart rate and breathing, measured in minutes/day. It involves movement that is more than sedentary behavior but does not reach the intensity level of moderate-to-vigorous physical activity (MVPA). Light physical activities are typically those that can be performed during daily tasks or leisurely pursuits and do not typically lead to significant sweating or increased breathing rate.The measure will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Actimetry records. Change from pre-intervention in Steps count at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The objective students levels of physical activity and sedentary behavior will be accessed through the actimetry recordings.The total number of steps count per day during the monitoring period, which provides a measure of ambulatory activity.
  The measure will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Actimetry records. Change from pre-intervention in energy expenditure at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The objective students levels of physical activity and sedentary behavior will be accessed through the actimetry recordings. Energy expenditure refers to the amount of energy, measured in calories or joules, that an individual uses or expands during a specific period of time.
  The measure will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Actimetry records. Change from pre-intervention in sedentary breaks at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The objective students levels of physical activity and sedentary behavior will be accessed through the actimetry recordings. Sedentary breaks refer to short periods of time during which individuals interrupt prolonged sitting or sedentary behavior by engaging in light physical activity or standing.
  The measure will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Actimetry records. Change from pre-intervention in Sedentary time at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The objective students levels of physical activity and sedentary behavior will be accessed through the actimetry recordings. The sedentary time is the total duration of sedentary behavior, defined as periods of minimal movement or activity, measured in minutes/day.
  The measure will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Actimetry records. Change from pre-intervention in prolonged sedentary bouts at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The objective students levels of physical activity and sedentary behavior will be accessed through the actimetry recordings. Prolonged sedentary bouts refer to extended periods of time during which individuals engage in minimal physical activity or remain in a seated or reclined position without interruption. These bouts typically last for prolonged durations, measured in minutes/day, often exceeding 30 minutes or more at a time.The measure will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Actimetry records. Change from pre-intervention in vector of the dynamic body acceleration (VeDBA) at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The objective students levels of physical activity and sedentary behavior will be accessed through the actimetry recordings. The VeDBA quantifies the dynamic acceleration of an body movements in three-dimensional space. The dynamic acceleration captured by the accelerometer reflects the intensity, accounting for both changes in speed and changes in direction. Researchers use VeDBA as a proxy for overall energy expenditure or activity levels in natural environments. Higher VeDBA values typically indicate more vigorous or energetic movements, while lower values suggest periods of rest or low activity.
  The measure will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Physical fitness markers - Strength. Change from pre-intervention in the force developed during a maximal isometric contraction of the quadriceps at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The students level of physical fitness will be assessed through a muscular strength test.
  The maximum isometric strength of the quadriceps during the strength test will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Physical fitness markers - Power. Change from pre-intervention in height of jump at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The squat jump is plyometric exercise in which a person bends their knees to lower their body into a squat position, then performs an explosive jump upwards by extending the hips, knees, and ankles simultaneously. During this exercise, the height of jump will be measured (in cm).
  The high of jump will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Physical fitness markers - Power. Change from pre-intervention in time of flight at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The students level of physical fitness will be assessed through a power test, a vertical jump. During this exercise, the time of flight will be measured (in seconds).
  The time of flight will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Physical fitness markers - Power. Change from pre-intervention in relative power at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The students level of physical fitness will be assessed through a power test, a vertical jump. During this exercise, the relative power can be estimated. The relative power will be done at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Physical fitness markers - Endurance. Change from pre-intervention in speed through the endurance test at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The students level of physical fitness will be assessed through a cardiorespiratory endurance test (modified VAMEVAL). The speed through the endurance will be recorded at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Physical fitness markers - Endurance. Change from pre-intervention in VO2max through the endurance test at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The students level of physical fitness will be assessed through a cardiorespiratory endurance test (modified VAMEVAL). During this test, the velocity at maximal aerobic (VMA) is the maximum speed (velocity) reached where the individual can still maintain aerobic metabolism without transitioning into anaerobic metabolism. VO2max refers to the maximum rate of oxygen consumption during intense exercise, typically measured in milliliters of oxygen per kilogram of body weight per minute (ml/kg/min). It is a key indicator of an individual's cardiovascular fitness and aerobic endurance. The VO2max was estimated as 3.5 times VMA. The VO2max through the endurance will be recorded at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Physical fitness markers - Endurance. Change from pre-intervention in heart rate during the endurance test at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The students level of physical fitness will be assessed through a cardiorespiratory endurance test (modified VAMEVAL). The heart rate will be measured at three moments: maximum, submaximal, at 1 minute, and 3 minutes of recovery. The measure will be recorded at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Body composition markers. Change from the pre-intervention in Body Mass Index (BMI) at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The BMI is a measure used to assess an individual's body weight in relation to their height. It's calculated by dividing a person's weight in kilograms by the square of their height in meters (BMI = weight in kilograms / (height in meters)²). BMI provides a general indication of whether a person's weight falls within a healthy range relative to their height. Here's how BMI categories are typically interpreted:
  Underweight: BMI less than 18.5 Normal weight: BMI between 18.5 and 24.9 Overweight: BMI between 25 and 29.9 Obesity: BMI 30 or greater
  The measure will be recorded at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Body composition markers. Change from the pre-intervention in fat mass at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The students body composition will be assessed using impedance metric variables.The fat mass metric represents the total amount of body fat. It's often expressed in kilograms or as a percentage of total body weight. The measure will be recorded at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Body composition markers. Change from the pre-intervention in Skeletal muscle mass at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The students body composition will be assessed using impedance metric variables. Skeletal muscle mass refers to the total mass or amount of skeletal muscle tissue in the body. It's often expressed in kilograms or as a percentage of total body weight.
  The measure will be recorded at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 Score)
Body composition markers.Change from the pre-intervention in total body hydration at the post-interventional measure at Week 27. | Week 1 (Pre-intervention) and Week 27 (Post-intervention)
  The students body composition will be assessed using impedance metric variables.The total body hydration metric represents the total amount of water present in the body, including intracellular and extracellular water compartments. It's often expressed in liters or as a percentage of total body weight. The measure will be recorded at different time frame:
  * Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  * Post-interventional measure at week 27 : after the modules (for the control and interventional groups).
  Change = (Week 27 score - Week 1 score)
Composite score - Student's satisfaction. Score ranging from 0 to 100 accessing the student's level of satisfaction of the stress module. | Week 9,11,10 - 16,17,18 - 24,25,26
  The composite score will be the mean of two sub-scores :
  1. A stress module specific score. Mean of the scores obtained at the three 100-mm VAS ranging from 0 (absolutely not) to 100 (completely) :
     * "Do you think the intervention has helped you to decrease your stress level?"
     * "Do you think the intervention allowed you to better manage the stressful events you encountered?"
  2. A stress module general score. Mean of the scores obtained at the 100-mm VAS ranging from 0 (absolutely not) to 100 (completely) :
     * "Do you think the proposed goals were suitable for your daily life?"
     * "Do you think you can sustain the habit changes?"
  Theses measures will be done at the session 3, i.e. approximately at week 9,11,10 for the first phase, at week 16,17,18 for the second phase and at week 24,25,26 for the third phase.
Composite score - Student's satisfaction. Score ranging from 0 to 100 accessing the student's level of satisfaction of the sedentary behaviors and physical activity module. | Week 9,11,10 - 16,17,18 - 24,25,26
  The composite score will be the mean of two sub-scores :
  1. A sedentary behaviors and physical activity module specific score. Mean of the scores obtained at the three 100-mm VAS ranging from 0 (absolutely not) to 100 (completely) :
     * "Do you think the module has helped you increase your level of physical fitness?")
     * "Do you think the module has helped you increase your level of physical activity?")
     * "Do you think the module has helped you decrease your level of sedentary behaviours?"
  2. A sedentary behaviors and physical activity module general score. Mean of the scores obtained at the two 100-mm VAS ranging from 0 (absolutely not) to 100 (completely) :
     * "Do you think the proposed goals were suitable for your daily life?"
     * "Do you think you can sustain the habit changes?"
  Theses measure will be done at the session 3, i.e. approximately at week 9,11,10 (1st phase), 16,17,18 (2n phase), 24,25,26 (3rd phase).
Composite score - Student's satisfaction. Score ranging from 0 to 100 accessing the student's level of satisfaction of the sleep module. | Week 9,11,10 - 16,17,18 - 24,25,26
  The composite score will be the mean of two sub-scores :
  1. A sleep module specific score. Mean of the scores obtained at the two 100-mm VAS ranging from 0 (absolutely not) to 100 (completely) :
     * "Do you think the module has helped you to improve your sleep?"
     * "Do you think the module has helped you to decrease your fatigue?"
  2. A sleep module general score. Mean of the scores obtained at the two 100-mm VAS ranging from 0 (absolutely not) to 100 (completely) :
     * "Do you think the proposed goals were suitable for your daily life?"
     * "Do you think you can sustain the habit changes?"
  Theses measure will be done at the session 3, i.e. approximately at week 9,11,10 for the first phase, at week 16,17,18 for the second phase and at week 24,25,26 for the third phase.
Question recommendation. Answer to the question "Would you recommend a friend to participate at the PROMESS project?" asked during the post-intervention. | Week 27 (Post-intervention)
  "Would you recommend a friend to participate in PROMESS?" The answer may be YES or NO. This will provide information on students' willingness to recommend the project and may represents their overall perception and appreciation of the project. This measure will be done during the post-interventional period at week 27 (for the control and interventional groups).
Question Habits change. Answer to the question "Do you think that your participation at the PROMESS project has modified your health behaviors/actions?" asked during the post-intervention. | Week 27 (Post-intervention)
  "Health behavior refers to all individual actions and habits that have an impact on health, including lifestyle choices, hygiene practices, diets, physical activity, sleep, use of substances such as tobacco and alcohol, stress management and compliance with medical recommendations. These behaviors play a crucial role in disease prevention, health promotion and overall well-being. Based on this definition, do you think that your participation at the PROMESS project has modified your health behaviors/actions?". The answer can be YES or NO.This measure will be done during the post-interventional period at week 27 (for the control and interventional groups).
Question Habits change. Answer to the question ""For which behaviors do you think you have modified your habits/actions?" asked during the post-intervention. | Week 27 (Post-intervention)
  If the student answers yes at the previous question ("Do you think that your participation at the PROMESS project has modified your health behaviors/actions?"), he/she will be asked: "For which behaviors do you think you have modified your habits/actions?". They may answer YES (positive changes), YES (negative change), NO (no change for this behavior) among a pre-established list of behaviors (stress, sleep, sedentary or physical activity behaviors). They may also declare additional different habits changes. This measure will be done during the post-interventional period at week 27 (for the control and interventional groups).

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Schlatter, Dr., Principal Investigator — RESHAPE U1290 INSERM UCBL-LYON 1 Rockfeller, Lyon France.
Locations (1):
- RESHAPE, Lyon, France

IPD SHARING:
Plan to Share IPD: No